CLINICAL TRIAL: NCT02791269
Title: Expanded Access Program of PEGASYS® (Peg Interferon Alpha-2a 40 KD) in Patients With HBeAg-Positive And HBeAg-Negative Chronic Hepatitis B
Brief Title: A Study of Peginterferon Alfa-2a in Participants With Chronic Hepatitis B Virus (HBV) in an Expanded Access Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19295
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (2):
- HBeAg Negative Participants (Experimental): HBeAg negative participants will receive peginterferon alfa-2a 180 micrograms (mcg) subcutaneous (SC) injection once weekly (QW) for 48 weeks followed by a 24 weeks treatment-free follow-up period.
  Interventions: Drug: Peginterferon alfa-2a
- HBeAg Positive Participants (Experimental): HBeAg Positive participants will receive peginterferon alfa-2a 180 mcg SC injection QW for 48 weeks followed by a 24 weeks treatment-free follow-up period.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180 mcg SC injection QW for 48 weeks.
  Other Names: Pegasys

SUMMARY:
This is an expanded access, multicenter, national, open-label, and non-randomized study to analyze the safety of peginterferon alfa-2a in participants with hepatitis B e antigen (HBeAg) positive and HBeAg negative chronic HBV infection. All participants will receive 48 weeks treatment of peginterferon alfa-2a monotherapy, followed by a 24 week treatment-free follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Non-cirrhotic participants
* Hepatitis B surface antigen (HBsAg) positive for at least 6 months
* Hepatitis B surface antibody (anti-HBs) negative
* Elevated serum alanine aminotransferase (ALT) greater than (>) upper limit of normal (ULN) but less than or equal to (</=) 10 times of ULN
* HBeAg positive participants: HBV DNA > 500,000 copies/mL, HBeAg negative participants: HBV DNA >100,000 copies/mL by polymerase chain reaction (PCR)
* Participants with chronic hepatitis B (CHB) who are treatment-naive
* No previous antiviral treatment with interferon (IFN: standard or pegylated) or with a nucleoside analogue
* For women of childbearing potential: negative urine or serum pregnancy test documented within the 24-hour period prior to the first dose of test drug. Willingness to use reliable contraception during the study and for 3 months after treatment completion

Exclusion Criteria:

* Previous antiviral or IFN-based therapy for CHB before enrolment
* Pregnant or breast feeding women participants
* Evidence of decompensated liver disease
* Co-infection with active hepatitis A, hepatitis C, hepatitis D and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis
* Previous or current hepatocellular carcinoma
* History of or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Alpha-fetoprotein levels of >100 nanograms (ng)/mL
* Severe psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the participant, in the opinion of the investigator, unsuitable for the study
* Thyroid disease uncontrolled by prescribed medications
* Evidence of severe retinopathy
* Alcohol intake more than 3 standard drinks per day for men and 2 standard drinks per day for women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- New Zealand (6):
  - Auckland
  - Hamilton
  - New Plymouth
  - Riccarton, Christchurch
  - Rotorua
  - Whangarei

RESULTS

PARTICIPANT FLOW:
Groups:
- HBeAg Negative Participants: Hepatitis B e antigen (HBeAg) negative participants received peginterferon alfa-2a 180 micrograms (mcg) subcutaneous (SC) injection once weekly (QW) for 48 weeks followed by a 24 weeks treatment-free follow-up period.
- HBeAg Positive Participants: HBeAg positive participants received peginterferon alfa-2a 180 mcg SC injection QW for 48 weeks followed by a 24 weeks treatment-free follow-up period.
Period: Overall Study
Arm/Group | HBeAg Negative Participants | HBeAg Positive Participants
Started | 4 | 20
Completed | 4 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included participants who received at least one dose of study medication and had one subsequent post baseline safety assessment.
Groups:
- HBeAg Negative Participants: HBeAg negative participants received peginterferon alfa-2a 180 mcg SC injection QW for 48 weeks followed by a 24 weeks treatment-free follow-up period.
- Total: Total of all reporting groups
Arm/Group | HBeAg Negative Participants | HBeAg Positive Participants | Total
Number analyzed (Participants) | 4 | 20 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.25 (5.75) | 31.57 (9.43) | 33.52 (9.88)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 4 | 13 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of HBeAg Positive Participants With Hepatitis B Virus-deoxy Ribonucleic Acid (HBV-DNA) Less Than (<) 100,000 Copies Per Milliliter (Copies/mL)
Description: HBV-DNA was assessed in plasma samples using quantitative Roche polymerase chain reaction (PCR) or Taqman tests.
Time Frame: End of 24-weeks follow-up (Week 72)
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of study medication and had one subsequent post baseline assessment. Here, "number of participants analyzed" signified those participants who were evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | HBeAg Positive Participants
Number analyzed (Participants) | 17
participants | 7

2. Primary Outcome: Number of Participants With HBV-DNA <20,000 Copies/mL
Description: HBV-DNA was assessed in plasma samples using quantitative Roche PCR or Taqman tests.
Time Frame: End of 24-weeks follow-up (Week 72)
Population: ITT population. Here, "number of participants analyzed" signified those participants who were evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | HBeAg Negative Participants | HBeAg Positive Participants
Number analyzed (Participants) | 3 | 17
participants | 0 | 3

3. Secondary Outcome: Number of Participants With HBV-DNA <400 Copies/mL
Description: HBV-DNA was assessed in plasma samples using quantitative Roche PCR or Taqman tests.
Time Frame: Week 48 (end of treatment) and Week 72 (end of follow-up)
Population: ITT population. Here, "number of participants analyzed" signified those participants who were evaluable for this outcome and "n" signified participants with evaluable data for a specified time point.
Measure: Number; unit: participants
Arm/Group | HBeAg Negative Participants | HBeAg Positive Participants
Number analyzed (Participants) | 4 | 18
participants
  Week 48 (n=4,18) | 3 | 6
  Week 72 (n=3,17) | 0 | 2

4. Secondary Outcome: Number of Participants With Hepatitis B Surface Antigen (HBsAg) Seroconversion
Description: HBsAg seroconversion was defined as the absence of HBsAg (a negative result for HBsAg) and the presence of anti-HBs (a positive result for anti-HBs). Both HBeAg positive and negative participants were HBsAg positive at baseline and absence of HBsAg (seroconversion) was analyzed.
Time Frame: Week 48 (end of treatment) and Week 72 (end of follow-up)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | HBeAg Negative Participants | HBeAg Positive Participants
Number analyzed (Participants) | 4 | 15
participants
  Week 48 (n=4,15) | 0 | 0
  Week 72 (n=4,13) | 0 | 0

5. Secondary Outcome: Number of Participants With Normalization of Alanine Aminotransferase (ALT) Level
Description: ALT is an enzyme found mainly in liver and is measured to check if the liver is damaged or diseased. In case of liver damage or disease, the liver releases ALT into the blood stream and the ALT level increases. Normal ALT level = less than upper limit of normal (40 units per liter).
Time Frame: Week 48 (end of treatment) and Week 72 (end of follow-up)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | HBeAg Negative Participants | HBeAg Positive Participants
Number analyzed (Participants) | 4 | 19
participants
  Week 48 (n=4,19) | 2 | 4
  Week 72 (n=4,17) | 4 | 7

6. Secondary Outcome: Number of Participants With HBeAg Seroconversion
Description: HBeAg seroconversion for HBeAg positive participants was defined as the loss of HBeAg (a negative result for HBeAg) and the presence of anti-HBe (a positive result for anti-HBe).
Time Frame: Week 48 (end of treatment) and Week 72 (end of follow-up)
Population: ITT population. Only HBeAg positive participants was planned to be reported. Here, "number of participants analyzed" signified those participants who were evaluable for this outcome and "n" signified participants with evaluable data for a specified time point.
Measure: Number; unit: participants
Arm/Group | HBeAg Positive Participants
Number analyzed (Participants) | 19
participants
  Week 48 (n=19) | 6
  Week 72 (n=17) | 6

ADVERSE EVENTS:
Time Frame: Baseline up to end of follow-up period (Approximately 72 weeks)
Description: Safety analysis population included participants who received at least one dose of study medication and had one subsequent post baseline safety assessment.
Arm/Group | HBeAg Negative Participants | HBeAg Positive Participants
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/20
Other Adverse Events (participants affected / at risk) | 3/4 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HBeAg Negative Participants (N=4) | HBeAg Positive Participants (N=20)
chest pain (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HBeAg Negative Participants (N=4) | HBeAg Positive Participants (N=20)
Depression (Nervous system disorders) | 2 | 1
Mood disturbance (Nervous system disorders) | 1 | 1
Tiredness (General disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Itchy skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Eye infection (Eye disorders) | 0 | 1
Non-productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blood in semen (Reproductive system and breast disorders) | 0 | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.